CLINICAL TRIAL: NCT02538510
Title: A Single Arm Phase I/II Study of MK-3475 Combined With Vorinostat for Recurrent Unresectable and/or Metastatic Squamous Cell Head and Neck Cancer and Recurrent Unresectable and/or Metastatic Salivary Gland Malignancies
Brief Title: Pembrolizumab and Vorinostat in Treating Patients With Recurrent Squamous Cell Head and Neck Cancer or Salivary Gland Cancer That Is Metastatic and/or Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Cristina Rodriguez, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9383; NCI-2015-01310 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MK-3475; 9383 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1715066 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2015-08-19; First posted 2015-09-02 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Recurrent Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Recurrent Nasopharynx Carcinoma; Recurrent Salivary Gland Carcinoma; Squamous Cell Carcinoma Metastatic in the Neck With Occult Primary; Stage III Major Salivary Gland Carcinoma; Stage III Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Stage III Nasopharyngeal Carcinoma; Stage IV Nasopharyngeal Carcinoma; Stage IVA Major Salivary Gland Carcinoma; Stage IVA Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Stage IVB Major Salivary Gland Carcinoma; Stage IVB Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Stage IVC Major Salivary Gland Carcinoma; Stage IVC Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Nasopharyngeal Neoplasms; Salivary Gland Neoplasms; Nasopharyngeal Carcinoma | interventions — pembrolizumab; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (vorinostat, pembrolizumab) (Experimental): Patients receive vorinostat PO QD or via PEG on days 1-5 and pembrolizumab IV over 30 minutes on day 1. Courses repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Drug: Vorinostat

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Vorinostat — Given PO or via PEG
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase I/II trial studies the side effects of pembrolizumab and vorinostat in treating patients with squamous cell head and neck cancer or salivary gland cancer that has come back, has spread to other places in the body and/or cannot be removed by surgery. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving pembrolizumab together with vorinostat may be a better treatment for head and neck cancer or salivary gland cancer.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive vorinostat orally (PO) once daily (QD) or via percutaneous endoscopic gastrostomy (PEG) on days 1-5 and pembrolizumab intravenously (IV) over 30 minutes on day 1. Courses repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and every 8-12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Phase I run in: biopsy proven RMHNSCC with the following primary sites: nasopharynx, paranasal sinus, nasal cavity, skin/cutaneous sites; patients with unknown head and neck primary sites will be enrolled; patients with recurrent or metastatic squamous cell carcinomas of the head and neck (regardless of primary site) who are either unwilling to receive or have contraindications (deemed by treating physician) to standard systemic chemotherapy will also be eligible; patients with biopsy proven RMSGC be eligible as well
* Phase II expansion: biopsy proven RMHNSCC, of any primary site (including unknown primary) and RMSGC will be eligible
* Have evidence of disease progression by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria within 3 months prior to study enrollment; if the patient was receiving a prior line of systemic therapy, he/she should have evidence of disease progression on that line of treatment prior to enrollment
* Have received any number lines of prior systemic therapy (including systemic therapy in the curative intent setting)
* Be willing and able to provide written informed consent for the trial and comply with the study visit requirements
* Have measurable disease based on RECIST 1.1
* Have provided tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L
* Serum creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated* creatinine clearance >= 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrC])

  * Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin =< 1.5 x ULN
* Aspartate aminotransferase (AST) (glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (glutamate pyruvate transaminase [SGPT]) =< 1.5 x ULN
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Patient is < 5 years free of another primary malignancy, except: a) if the other malignancy is basal cell carcinoma or cervical carcinoma in situ or b) if the other primary malignancy is not considered clinically significant and is requiring no active intervention
* SECOND COURSE PHASE (RETREATMENT PERIOD FOR POST-COMPLETE RESPONSE RELAPSE ONLY)
* Subjects may be eligible to receive MK-3475 in the second course phase of this study if the study remains open and the subject meets the following conditions:
* Stopped initial treatment with MK-3475 after attaining an investigator-determined confirmed response according to RECIST1.1 response criteria
* Was treated for at least 24 weeks with MK-3475 before discontinuing therapy
* Received at least four treatments with MK-3475 beyond the date when the initial complete response (CR) was declared
* Experienced an investigator-determined confirmed cutaneous or radiographic disease progression after stopping their initial treatment with MK-3475
* Did not receive any anti-cancer treatment since the last dose of MK-3475
* Have a performance status of 0 or 1 on the ECOG performance scale
* Demonstrate adequate organ function as detailed above
* Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving retreatment with study medication
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of child bearing potential are those who have not been surgically sterilized or have not been free from menses for > 2 year; male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Does not have a history or current evidence of any condition, therapy, or laboratory abnormality that might interfere with the subject's participation for the full duration of the trial or is not in the best interest of the subject to participate, in the opinion of the treating investigator

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has had a prior monoclonal antibody within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study; subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-programmed cell death 1 (PD-1), PD-L1, anti-programmed cell death ligand 2 (PD-L2), anti-cluster of differentiation (CD)137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways); patients who have previously received MK-3475 or participated in an MK-3475 clinical trial will be ineligible
* Has received prior therapy with vorinostat or other epigenetic agent
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B virus surface antigen [HBsAg] reactive) or hepatitis C (HCV) (e.g., HCV RNA [ribonucleic acid] qualitative is detected)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment
* Requires total parenteral nutrition and is unable to swallow pills or unable to take a suspension through a gastrostomy tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10-08 (Actual); Primary Completion 2019-09-28 (Actual); Study Completion 2023-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Rodriguez, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Pan C, Wu QV, Voutsinas J, Houlton JJ, Barber B, Futran N, Laramore GE, Liao JJ, Parvathaneni U, Martins RG, Fromm JR, Rodriguez CP. Neutrophil to lymphocyte ratio and peripheral blood biomarkers correlate with survival outcomes but not response among head and neck and salivary cancer treated with pembrolizumab and vorinostat. Head Neck. 2023 Feb;45(2):391-397. doi: 10.1002/hed.27252. Epub 2022 Nov 22. PMID 36412064
- [Derived] Rodriguez CP, Wu QV, Voutsinas J, Fromm JR, Jiang X, Pillarisetty VG, Lee SM, Santana-Davila R, Goulart B, Baik CS, Chow LQM, Eaton K, Martins R. A Phase II Trial of Pembrolizumab and Vorinostat in Recurrent Metastatic Head and Neck Squamous Cell Carcinomas and Salivary Gland Cancer. Clin Cancer Res. 2020 Feb 15;26(4):837-845. doi: 10.1158/1078-0432.CCR-19-2214. Epub 2019 Dec 3. PMID 31796519

RESULTS

PARTICIPANT FLOW:
Groups:
- Head and Neck Squamous Cell Carcinoma: MK-3475 combined with vorinostat,HNSCC patients
- Salivary Gland Carcinoma: MK-3475 combined with votinostat, SGC patients
Period: Overall Study
Arm/Group | Head and Neck Squamous Cell Carcinoma | Salivary Gland Carcinoma
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: RMHNSCC with the following primary sites:nasopharynx, paranasal sinus, nasal cavity, skin/cutaneous sites. Pts with unknown HN primary sites will be enrolled. Patients with biopsy proven RMSGC be eligible as well
Groups:
- Head and Neck Squamous Cell Carcinoma: Head and Neck Squamous Cell Carcinoma patients
- Salivary Gland Carcinoma: Salivary Gland Carcinoma patients
- Total: Total of all reporting groups
Arm/Group | Head and Neck Squamous Cell Carcinoma | Salivary Gland Carcinoma | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 18 | 32
  >=65 years | 11 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.12 (8.99) | 56.84 (13.64) | 59.98 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 11
  Male | 23 | 16 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 24 | 24 | 48
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 20 | 21 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Toxicity Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: Toxicities will be summarized as the number and percentage of patients with each type of toxicity, per Criteria for Adverse Events version 4.0
Time Frame: Up to 30 days after the completion of study treatment
Population: Only G3 toxicities and toxicities requiring dose hold/reduction recorded.
Measure: Count of Participants; unit: Participants
Groups:
- Head and Neck Squamous Cell Carcinoma: AEs experienced with MK-3475 combined with vorinostat in HNSCC patients
- Salivary Gland Carcinoma: AEs experienced with MK-3475 combined with vorinostat in salivary gland carcinoma patients
Arm/Group | Head and Neck Squamous Cell Carcinoma | Salivary Gland Carcinoma
Number analyzed (Participants) | 25 | 25
Participants
  Adrenal insufficiency | 1 | 1
  ALT increase | 0 | 1
  Anorexia | 0 | 1
  Arthiritis | 0 | 1
  AST increase | 0 | 1
  Cough | 1 | 0
  Increased Creatinine | 2 | 5
  Dermatitis | 1 | 0
  Diarrhea | 0 | 1
  Fever with leukocytosis | 0 | 1
  Fatigue | 2 | 4
  Hyponatremia | 2 | 0
  Hypothyroidism | 1 | 0
  Colitis and Ileitis | 1 | 0
  Malaise | 1 | 0
  Nausea | 1 | 3
  Nephritis | 0 | 1
  Pneumonitis | 1 | 0
  Neuritis | 0 | 1
  Tracheitis/Epiglottitis | 1 | 0
  Vomiting | 1 | 2

2. Secondary Outcome: Objective Response Rate
Description: Radiologic assessments of measurable disease will be performed using radiographic imaging. RECIST 1.1 and immune response criteria will be used to assess response to therapy. Responses will be summarized as frequencies and percentages.
Time Frame: Up to 2 years
Population: 6 patients were not evaluated as they did not have at least 1 set of follow up scans while on study, (N=2 salivary patients, N=4 SCC patients)
Measure: Count of Participants; unit: Participants
Groups:
- Head and Neck Squamous Cell: Head and Neck Squamous Cell RECIST 1.1
- Salivary Gland Carcinoma: RECIST 1.1 response rate salivary gland
Arm/Group | Head and Neck Squamous Cell | Salivary Gland Carcinoma
Number analyzed (Participants) | 21 | 23
Participants
  partial response | 8 | 4
  stable disease | 8 | 13
  progressive disease | 5 | 6

3. Secondary Outcome: Overall Survival
Description: The Kaplan Meier methods will be used to estimate overall survival.
Time Frame: Up to 7 years 6 months
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Head and Neck Squamous Cell Carcinoma | Salivary Gland Carcinoma
Number analyzed (Participants) | 25 | 25
Months | 23.2 [12.9 to 33.5] | 28.04 [17.8 to 38.3]

4. Secondary Outcome: Progression Free Survival
Description: The Kaplan Meier methods will be used to estimate progression free survival.
Time Frame: Up to 2 years
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Head and Neck Squamous Cell Carcinoma | Salivary Gland Carcinoma
Number analyzed (Participants) | 25 | 25
Months | 12.6 [8.1 to 15.3] | 14.0 [8.5 to 24.5]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored for up to 7 years and 6 months; serious and/or other adverse events were assessed up to 3 years and 6 months.
Description: Adverse events are collected from the first dose of Mk-3475 or Vorinostat, and are collected through 30 days post the last dose of therapy.
Groups:
- Head and Neck Squamous Cell Carcinoma: MK-3475 combined with vorinostat in HNSCC patients
- Salivary Gland Carcinoma: MK-3475 combined with vorinostat in SGC patients
Arm/Group | Head and Neck Squamous Cell Carcinoma | Salivary Gland Carcinoma
All-Cause Mortality (participants affected / at risk) | 22/25 | 23/25
Serious Adverse Events (participants affected / at risk) | 1/25 | 1/25
Other Adverse Events (participants affected / at risk) | 11/25 | 19/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Head and Neck Squamous Cell Carcinoma (N=25) | Salivary Gland Carcinoma (N=25)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Head and Neck Squamous Cell Carcinoma (N=25) | Salivary Gland Carcinoma (N=25)
alanine amintotransferase (ALT) increased (Hepatobiliary disorders) | 0 (0) | 1 (1)
asparate aminotransferase (AST) increased (Hepatobiliary disorders) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
creatinine increased (Renal and urinary disorders) | 2 (2) | 5 (6)
Fatigue (General disorders) | 2 (3) | 4 (6)
Fever with Leukocytosis (Infections and infestations) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Immune system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT02538510/Prot_SAP_000.pdf